CLINICAL TRIAL: NCT01411800
Title: A Phase 1, Randomized, Open-Label, Two-Way Crossover Study of Two Oral Formulations of LX1033 in Healthy Human Subjects
Brief Title: An Open-Label Study of Two Formulations of LX1033 in Healthy Human Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Lexicon Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LX1033.1-103-NRM; LX1033.103 (Other: Lexicon Pharmaceuticals, Inc.)
Record Dates: First submitted 2011-08-05; First posted 2011-08-08 (Estimated); Last update posted 2012-07-20 (Estimated); Status verified 2012-07

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment A (Experimental): 500 mg LX1033, capsules administered two times per day orally
  Interventions: Drug: 250 mg capsule
- Treatment B (Experimental): 500 mg LX1033, tablets administered two times per day orally
  Interventions: Drug: 250 mg tablets

INTERVENTIONS:
Drug: 250 mg capsule — Two 250 mg capsules will be administered for 500 mg dose
  Arms: Treatment A
Drug: 250 mg tablets — Two 250 mg tablets will be administered for a 500 mg dose
  Arms: Treatment B

SUMMARY:
The purpose of this study is to assess the pharmacodynamic effects, pharmacokinetics, and safety of two oral formulations (tablet and capsule) of LX1033 in normal healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects age 18 to 55 years
* Vital signs acceptable at Screening
* Body mass index (BMI) between 18 and 35 kg/m^2 at Screening
* Considered to be in good health, as determined by the Investigator
* Normal ECG findings
* Negative urine screen for drugs of abuse and negative breath test for alcohol
* Negative hepatitis B surface antigen, hepatitis C antibody, and HIV1 and HIV2 antibody tests within the last 28 days
* Ability to provide written informed consent

Exclusion Criteria:

* Use of any medication (including acetaminophen) within 5 days of dosing
* Use of any investigational agent or selective serotonin reuptake inhibitors (SSRIs) within 30 days of study start
* Administration of any protein or antibodies within 90 days of study start
* Donation or loss of greater than 450 mL of blood within 45 days of study start
* Known history of hepatic disease or significantly abnormal liver function tests
* History of alcoholism or substance abuse within 3 years prior to study start
* Participation in any other clinical study within 30 days preceding the first dose of study drug
* Positive serum pregnancy test

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2011-08; Primary Completion 2011-10 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Urinary 5-HIAA levels | 34 days
Plasma 5-HIAA levels | 30 days

SECONDARY OUTCOMES:
Maximum observed plasma concentration | 32 days
Time at which maximum observed plasma concentration occurs | 32 days
Half-life of the drug in plasma | 32 days

CONTACTS AND LOCATIONS:
Overall Officials: Ikenna Ogbaa, MD, Study Director — Lexicon Pharmaceuticals, Inc.
Locations (1):
- Lexicon Investigational Site, Overland Park, Kansas, United States